CLINICAL TRIAL: NCT06390696
Title: Biodiversity Interventions for Well-being - the Effect of Biodiversity Exposure on Atopic Dermatitis
Brief Title: Sand Play - the Effect of Biodiversity Exposure on Atopic Dermatitis
Acronym: BIWE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Natural Resources Institute Finland (Other Government)
Collaborators: Tampere University (Other)
Responsible Party: Principal Investigator, Aki Sinkkonen, Lead Researcher, Natural Resources Institute Finland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R22127
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Atopic Dermatitis; Nature, Human; Microbial Colonization; Immune System and Related Disorders
Keywords: Atopy; Biodiversity; Commensal microbiota; Microbial exposure
MeSH Terms: conditions — Dermatitis, Atopic; Communicable Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microbial intervention (Experimental): Children receive an indoor sandbox and cultivation set including soil- and plant-based material with high microbial diversity.
  Interventions: Biological: Microbial intervention
- placebo (Placebo Comparator): Children receive an indoor sandbox and cultivation set including placebo material with low microbial diversity.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Microbial intervention — Children in microbial intervention arm receive an indoor sandbox containing play sand enriched with organic leaf compost, moss and humus substances. Families also receive an indoor cultivation set including growing box, seeds, spray bottle, plant lamp and microbe rich growing medium containing organic leaf compost, moss, biochar and humus substances.
  Arms: Microbial intervention
Other: Placebo — Children in placebo arm receive an indoor sandbox containing visually similar play sand modified with peat with low microbial diversity. Families also receive an indoor cultivation set including growing box, seeds, spray bottle, plant lamp and growing medium containing peat, inorganic fertilizers, and potting gravel with low microbial diversity.
  Arms: placebo

SUMMARY:
The prevalence of atopic dermatitis has increased along with urbanization and biodiversity loss. According to biodiversity hypothesis, the main reason is urban lifestyle and reduced contact to microbial diversity. Previous studies indicate association between atopic dermatitis and exposure to natural microbes in childhood.

Sand Play - the Effect of Biodiversity Exposure on Atopic Dermatitis will investigate whether the exposure to microbial diversity in sandbox reduces the symptoms of atopic dermatitis, alters commensal microbiota and modifies immune regulation in children.

DETAILED DESCRIPTION:
Our specific aims are:

To assess if exposure to microbial diversity reduces Eczema Area and Severity Index (EASI) and Patient-Oriented Eczema Measure (POEM).

Assess whether the sand play alters plasma cytokine profiles, white blood cell distributions, allergy specific IgE, and commensal microbial communities on skin, in saliva and gut.

The investigators will recruit approximately 80 (40 study subjects per treatment) subjects with atopic dermatitis and aged between 2-5.

ELIGIBILITY:
Inclusion Criteria:

* Eczema Area and Severity Index ≥ 2

Exclusion Criteria:

* Eczema Area and Severity Index < 2
* Immune deficiencies, i.e., antibody deficiency
* Immunosuppressive systematic medications
* A disease affecting immune response (e.g., colitis ulcerosa, rheumatoid arthritis, Crohn's disease, diabetes)
* Cancer diagnosis
* Topical medication for the treatment of atopic dermatitis during the trial
* Disability affecting the immune response (e.g. Down's syndrome)
* Non-participation in the national vaccine program
* Participation in another intervention or follow-up study

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Eczema Area and Severity Index (EASI) | Baseline, 2 month, 6 month
  EASI reduced by at least 50% from baseline in microbial intervention treatment. The minimum EASI score is 0 and the maximum EASI score is 72.

SECONDARY OUTCOMES:
The Patient-Oriented Eczema Measure | Baseline, 2 month, 6 month
  Lower score on the Patient-Oriented Eczema Measure (POEM) among microbial intervention arm compared to placebo arm after intervention. The total POEM score can range from 0 to 28, with higher scores indicating more severe eczema symptoms.
Allergy specific Immunoglobulin E | Baseline, 2 month, 6 month
  It will be analyzed if allergy specific IgE is different between treatments
Plasma cytokines | Baseline, 2 month, 6 month
  Cytokines will be analyzed analyzed with Meso Scale.
Distribution of white blood cells | Baseline, 2 month, 6 month
  It will be analyzed if the distribution is different between treatments
Skin microbiota | Baseline, 2 month, 6 month
  It will be analyzed if skin microbial communities are different between treatments
Saliva microbiota | Baseline, 2 month, 6 month
  It will be analyzed if saliva microbial communities are different between treatments
Gut microbiota | Baseline, 2 month, 6 month
  It will be analyzed if stool microbial communities are different between treatments
Infectious diseases | Baseline, 2 month, 6 month
  Infections will be recorded with questionnaires.
Perceived Stress Scale | Baseline, 2 month, 6 month
  Lower score on a perceived stress scale among guardians in intervention arm compared to placebo arm that indicates lower perceived stress levels among guardians in intervention arm. Minimum 0, maximum 40.
Warwick-Edinburgh Mental Wellbeing Scale | Baseline, 2 month, 6 month
  Higher score on a Warwick-Edinburhg Mental Wellbeing scale among guardians in intervention arm compared to placebo arm that indicates better mental well-being among guardians in intervention arm. Minimum 14, maximum 70.
Depression Scale | Baseline, 2 month, 6 month
  Lower score on a Depression scale among guardians in intervention arm compared to placebo arm that indicates lower levels of depression symptoms among guardians in intervention arm. Minimum 0, maximum 60.
Nature Relatedness Scale | Baseline, 2 month, 6 month
  Higher score on a Nature Relatedness scale among guardians in intervention arm compared to placebo arm that indicates stronger sense of connectedness to nature among intervention arm. Minimum 6, maximum 30.

OTHER OUTCOMES:
Association between atopic dermatitis and skin microbiota. | Baseline, 2 month, 6 month
  It will be assessed if changes in skin microbiota are associated with Eczema Area and Severity Index and the Patient-Oriented Eczema Measure.
Association between commensal microbiota and other outcomes. | Baseline, 2 month, 6 month
  It will be assessed if commensal microbiota on skin, saliva or gut are associated with plasma cytokines, IgE or white blood cell distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Aki Sinkkonen, Principal Investigator — Natural Resources Institute Finland
Locations (2):
- Finland (2):
  - Natural Resources Institute Finland, Helsinki, Uusimaa
  - Tampere University, Tampere